CLINICAL TRIAL: NCT01387763
Title: Danish Study of Low-dose Interferon Alpha Versus Hydroxyurea in the Treatment of Philadelphia Chromosome Negative (Ph-)Chronic Myeloid Neoplasms.
Brief Title: A Study of Low Dose Interferon Alpha Versus Hydroxyurea in Treatment of Chronic Myeloid Neoplasms
Acronym: DALIAH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Stauffer Larsen (Other)
Responsible Party: Sponsor-Investigator, Thomas Stauffer Larsen, MD PhD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: daliah2011
Record Dates: First submitted 2011-06-23; First posted 2011-07-06 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia; Primary Myelofibrosis
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis | interventions — peginterferon alfa-2b; peginterferon alfa-2a; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- PegIntron <= 60 years (Active Comparator): In patients <= 60 years PegIntron is started at low-dose 35 micrograms once weekly. Dose escalation to 50 micrograms weekly if lack of complete hematological response at 4 months or lack of at least partial molecular response at 8 months. If complete hematological response or lack of at least partial molecular response is not achieved at 50 micrograms weekly at 12 months and 18 months respectively, dose escalation to 96 micrograms weekly.
  Interventions: Drug: PegIntron
- Pegasys <= 60 years (Active Comparator): In patients <= 60 years Pegasys is started at low-dose 45 micrograms once weekly. Dose escalation to 90 micrograms weekly if lack of complete hematological response at 4 months or lack of at least partial molecular response at 8 months. If complete hematological response or lack of at least partial molecular response is not achieved at 90 micrograms weekly at 12 months and 18 months respectively, dose escalation to 135 micrograms weekly.
  Interventions: Drug: Pegasys
- PegIntron > 60 years (Active Comparator): In patients < 60 years PegIntron is started at low-dose 35 micrograms once weekly. Dose escalation to 50 micrograms weekly if lack of complete hematological response at 4 months or lack of at least partial molecular response at 8 months. If complete hematological response or lack of at least partial molecular response is not achieved at 50 micrograms weekly at 12 months and 18 months respectively, dose escalation to 96 micrograms weekly.
  Interventions: Drug: PegIntron
- Pegasys > 60 years (Active Comparator): In patients > 60 years Pegasys is started at low-dose 45 micrograms once weekly. Dose escalation to 90 micrograms weekly if lack of complete hematological response at 4 months or lack of at least partial molecular response at 8 months. If complete hematological response or lack of at least partial molecular response is not achieved at 90 micrograms weekly at 12 months and 18 months respectively, dose escalation to 135 micrograms weekly.
  Interventions: Drug: Pegasys
- Hydroxyurea > 60 years (Active Comparator): Capsule Hydrea 500-2000 mg orally QD or BID
  Interventions: Drug: Hydrea

INTERVENTIONS:
Drug: PegIntron — PegIntron, prefilled syringe 50 micrograms/0.5 ml. 30 micrograms subcutaneously once weekly.
  Other Names: Pegylated interferon alpha 2b
  Arms: PegIntron <= 60 years
Drug: Pegasys — Pegasys, prefilled syringe 180 micrograms/0.5 ml 45 micrograms subcutaneously once weekly
  Other Names: Pegylated interferon alpha 2a
  Arms: Pegasys <= 60 years
Drug: PegIntron — PegIntron, prefilled syringe 50 micrograms/0.5 ml. 30 micrograms subcutaneously once weekly.
  Other Names: Pegylated interferon alpha 2b
  Arms: PegIntron > 60 years
Drug: Pegasys — Pegasys, prefilled syringe 180 micrograms/0.5 ml 45 micrograms subcutaneously once weekly
  Other Names: Pegylated interferon alpha 2a
  Arms: Pegasys > 60 years
Drug: Hydrea — Capsule Hydrea 500-2000 mg orally QD or BID
  Other Names: hydroxyurea; hydroxycarbamide
  Arms: Hydroxyurea > 60 years

SUMMARY:
The purpose of the study is to compare the efficacy and toxicity including quality of life of two types of low-dose interferon alpha compounds (PegIntron and Pegasys) with hydroxyurea (Hydrea), and to investigate the occurence of neutralizing antibodies against recombinant interferon.

DETAILED DESCRIPTION:
Chronic myeloid neoplasms (CMPN) consists of three main entities, polycythemia vera (PV), essential thrombocythemia (ET) and primary myelofibrosis (PMF). These three disorders have many overlapping clinical features. The diseases are clonal stem cell disorders characterized by a chronic excess production of mainly mature myeloid cells. The excess production of clonal red cells (in PV), platelets (in PV, ET and PMF) and leukocytes (mainly PV and PMF)leads to a highly increased risk of thrombosis. Patients may also suffer from constitutional symptoms, pruritus and splenomegaly. An inherent feature of these diseases are the risk of ET and PV of transformation to myelofibrosis and a risk of both ET, PV and PMF of leukemic transformation.

In 2005 major breakthrough in our understanding of the molecular pathophysiology was achieved with the identification of the JAK2 V617F mutation which is present in almost all patients with PV (98%) and about half of patients with ET and PMF. This somatic gain-of-function point mutation in the JAK2 tyrosine kinase leads to constitutive activation of the kinase. By this mechanism a clonal non-growth factor dependent myeloproliferation is established.

Traditionally the excess platelet and white cell production in ET, PV and PMF has been treated with cytoreductive agents such as hydroxyurea and busulfan in order to normalize the blood counts and thereby reducing the risk of thrombosis. However, in younger patients there is a concern of the leukemogenic potential of these agents. In younger patients an alternative treatment option is recombinant pegylated interferon alpha (IFN-alpha), which has demonstrated high clinical efficacy and has no leukemogenic potential. Within recent years IFN-alpha has demonstrated a capacity of inducing deep molecular remission (evaluated by JAK2 V617F qPCR) and normalisation of bone marrow morphology. These remissions have been sustained for up to 3 years after discontinuation of IFN-alpha therapy. Accordingly a perspective of changing the natural history of these disorders towards myelofibrosis and ultimately acute leukemia has emerged. However toxicity has been a major issue and drop-of rates have been reported consistently around 25 %.

It is well known from other diseases (e.g multiple sclerosis and hepatitis) that some patients develop neutralizing antibodies against IFN-alpha. This issue is however only scarcely investigated in CMPN and has never been tested in a prospective design.

The purpose of this study is to compare the efficacy (hematological and molecular) and toxicity profile of two different recombinant interferon alpha products, IFN-alpha2a and IFN-alpha2b in a prospective randomized design. In patients over the age of 60 there will be a third study arm with hydroxyurea.

In order to decrease drop out rates and thereby increasing response rates patients will be started of at a low-dose of IFN-alpha. If patients fail to respond or looses their response and develops neutralizing antibodies against IFN-alpha therapy will be stopped. If patients have a sustained deep molecular response (below 1 % JAK2 V617F mutated alleles for 12 months) therapy will be stopped to asses the sustainability of the remission off therapy.Patients over the age of 75 and intolerant or resistant to hydroxyurea will be offered rescue treatment with orally busulfan (Myleran). As an important part of the study quality of life will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years of age
* Newly diagnosed, or previously diagnosed untreated patients with ET, PV or PMF including prefibrotic myelofibrosis according to the WHO classification
* Active disease defined by one of the following criteria:
* need for phlebotomy
* leukocytosis > 10 mia/l
* thrombocytosis > 400 mia/l
* constitutional symptoms (fatigue, weight loss, night sweats or fewer > 38 degrees celsius)
* Pruritus
* splenomegaly causing symptoms
* previous thrombosis

Exclusion Criteria:

* Fertile women without a negative pregnancy test
* Other malignant disease within last 5 years
* ECOG performance score >/= 3
* Creatinine > 2x ULN
* Bilirubin > 1.5x ULN
* ALAT > 3x ULN
* Previous psychiatric disorder (depression)
* active autoimmune disease
* Uncontrolled thyroid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2012-01; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
molecular response (changes from baseline) | 18, 36 and 60 months
  Molecular responses (JAK V617F allele burden) are assessed by qPCR according to the ELN guidelines.

SECONDARY OUTCOMES:
toxicity (discontinuation of therapy due to intolerability) | 18 months
  The proportion of patients treated with PegIntron, Pegasys and Hydrea who need to discontinue therapy due to intolerability
Quality of life (changes from baseline) | 4, 12, 24, 36, 48 and 60 months
  Quality of life will be evaluated according to EORTC QLQ C-30 and MPN-SAF
Histopathological response (changes from baseline) | 36 and 60 months
  A bone marrow sample will be evaluated in order to detect and grade changes in bone marrow morphology.
Sustained molecular response (changes from level at time of discontinuation of therapy) | 12, 24 and 36 months
  investigation of the sustainability of an obtained molecular remission (<
  1% JAK2V617F mutated alleles) after discontinuation of interferon- alpha( Pegasys, PegIntron, Multiferon) or Hydrea.
Neutralizing antibodies against PegIntron and Pegasys | 24 months
  Proportion of patients treated with Peintron and Pegasys who have developed neutralizing antibodies.
hematological response | 12 months
  Hematological response will be evaluated according to the ELN guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas S Larsen, MD PhD, Principal Investigator — Dept. of Hematology, Odense University Hospital
Locations (8):
- Denmark (8):
  - Dept of Hematology, Aalborg hospital, Aalborg
  - Dept. of Hematology, Aarhus University Hospital, Aarhus
  - Dept of Hematology, Rigshospitalet, Copenhagen
  - Dept of Hematology, Esbjerg Hospital, Esbjerg
  - Dept of Hematology, Herlev Hospital, Herlev
  - Dept of Hematology, Holstebro Hospital, Holstebro
  - Dept of hematology, Odense University Hospital, Odense
  - Dept. of Hematology, Roskilde Hospital, Roskilde